CLINICAL TRIAL: NCT05741996
Title: Do Taping and Orthosis Affect Pain, Gait, or Functionality in Mild Knee Osteoarthritis? A Randomized Clinical Trial
Brief Title: Do Taping and Orthosis Affect Pain, Gait, or Functionality in Mild Knee Osteoarthritis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tezel Yıldırım Şahan, Clinical Researcher, Hacettepe University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-01
Record Dates: First submitted 2023-02-02; First posted 2023-02-23 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee
Keywords: knee osteoarthritis; athletic tape; brace; kinesiotape; gait
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Braces

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effetcs of Taping type and Orthosis on Pain, (Experimental): The order of the elastic taping, rigid taping, and braces was randomized using a computer-generated random sequence created before the research (Random.org). Both knees of each participant were taped and braced. The participants were allowed to become accustomed to the applied elastic taping, rigid taping, and braces before the gait analysis and evaluations. All the taping techniques and braces were similar for all the participants. The participants performed four evaluation condition trials at baseline and with the elastic taping, rigid taping, and braces after 45 minutes.
  Interventions: Behavioral: Taping
- Effetcs of Taping type and Orthosis on Gait and functionality (Experimental): The Western Ontario and McMaster Universities Turkish Version 3.1 (WOMAC) index is a self-administered questionnaire that assesses three aspects of a patient's health status -pain, stiffness, and physical function - in those with lower limb Osteoarthritis.
  Gait analysis was conducted using a 3-dimensional VICON gait analysis system (Workstation Version 4.0, Oxford, UK). Each participant was assessed four times before and after the applications.
  Interventions: Behavioral: Taping

INTERVENTIONS:
Behavioral: Taping — Taping types and brace acute effects for knee osteoartritis
  Other Names: Brace

SUMMARY:
Objective: The aim of this study was to compare the effects of elastic taping, rigid taping, and braces applied to women with mild knee Osteoartritis(OA) on pain, gait, and knee functionality.

Methods: This randomised study included 21 female patients (mean age of 53.81±6.20 years) with bilateral grade 2 knee OA according to the Kellgren & Lawrence Classification. Pain was evaluated with the visual analog scale, functionality was evaluated with the Western Ontario McMaster Osteoarthritis Index, and the kinetic, kinematic, and spatiotemporal parameters were evaluated using a three-dimensional gait analysis system at baseline (no application) and immediately after the application of elastic taping, rigid taping, and orthoses. The dependent variables were measured after 45 minute the application of four different conditions neutral, elastic taping, rigid taping, and knee brace on each participant with 1-day intervals.

DETAILED DESCRIPTION:
Objective: The aim of this study was to compare the effects of elastic taping, rigid taping, and braces applied to women with mild knee OA on pain, gait, and knee functionality.

Methods: This randomised study included 21 female patients (mean age of 53.81±6.20 years) with bilateral grade 2 knee OA according to the Kellgren & Lawrence Classification. Pain was evaluated with the visual analog scale, functionality was evaluated with the Western Ontario McMaster Osteoarthritis Index, and the kinetic, kinematic, and spatiotemporal parameters were evaluated using a three-dimensional gait analysis system at baseline (no application) and immediately after the application of elastic taping, rigid taping, and orthoses. The dependent variables were measured after 45 minute the application of four different conditions neutral, elastic taping, rigid taping, and knee brace on each participant with 1-day intervals.

ELIGIBILITY:
Inclusion Criteria:

* bilateral knee OA according to the criteria of the American College of Rheumatology
* had radiographically phase 2 based on the criteria identified by Kellgren & Lawrence

  -, had active knee pain
* did not receive any knee treatment in the last year
* could understand test and evaluations

Exclusion Criteria:

* experienced lower extremity trauma or underwent surgery
* had phase 3-4 Osteoarthritis
* had any orthopedic or neurologic problem affecting walking
* were allergic to taping
* did not walk independently on their own

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 21 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Pain Maasurements | 5 minute
  effects of them on pain

SECONDARY OUTCOMES:
Gait Measurements, Functionality Measurement | 10 minute
  effects of them on gait and functionality

CONTACTS AND LOCATIONS:
Overall Officials: Tezel Y Şahan, pHD, Principal Investigator — University of Health science
Locations (2):
- Turkey (Türkiye) (2):
  - Tezel Yıldırım Şahan, Ankara
  - University of Health Science, Ankara

IPD SHARING:
Plan to Share IPD: No
If they want from corresponding author then can be shaberable.

REFERENCES:
- [Result] Anvar N, Matlabi H, Safaiyan A, Allahverdipour H, Kolahi S. Effectiveness of self-management program on arthritis symptoms among older women: A randomized controlled trial study. Health Care Women Int. 2018 Dec;39(12):1326-1339. doi: 10.1080/07399332.2018.1438438. Epub 2018 Mar 5. PMID 29419362
- [Result] DeVita P, Aaboe J, Bartholdy C, Leonardis JM, Bliddal H, Henriksen M. Quadriceps-strengthening exercise and quadriceps and knee biomechanics during walking in knee osteoarthritis: A two-centre randomized controlled trial. Clin Biomech (Bristol). 2018 Nov;59:199-206. doi: 10.1016/j.clinbiomech.2018.09.016. Epub 2018 Sep 15. PMID 30273922
- [Result] Teo PL, Hinman RS, Egerton T, Dziedzic KS, Bennell KL. Identifying and Prioritizing Clinical Guideline Recommendations Most Relevant to Physical Therapy Practice for Hip and/or Knee Osteoarthritis. J Orthop Sports Phys Ther. 2019 Jul;49(7):501-512. doi: 10.2519/jospt.2019.8676. PMID 31258044